CLINICAL TRIAL: NCT01834430
Title: Effects of Delayed Enteral Nutrition on Inflammatory Responses and Immune Function Competence in Critically Ill Patients With Prolonged Fasting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing PLA General Hospital (Other)
Responsible Party: Principal Investigator, Gao Tao, Clinical Professor, Nanjing PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009NLY059
Record Dates: First submitted 2013-04-07; First posted 2013-04-17 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Severe Acute Pancreatitis Patients; Duodenal Fistula; Inflammatory Intestinal Obstruction
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- EN group (Experimental): The EN group gradually restored enteral nutrition, while the PN group continued to receive parenteral nutrition treatment. Both groups received between 20 to 25 kcal/kg/day and 1.5 g/kg/day of protein. Because of the low volume, concentration, and calorie amount, on the first day, tube feeding utilized 500 ml with the speed of 30 ~ 50 ml/h. On the second day, tube feeding utilized 1000 ml with the speed of 60 ~ 80 ml/h. On the third day, tube feeding utilized 1500 ~ 2000 ml with the speed of 100 ~ 120 ml/h. If enteral nutrition could not meet a patient's caloric requirements, PN supplement was started on the fourth day. The required calories and protein for each individual in the two groups was assumed to be achieved after three days of therapy. The PN group continued to receive parenteral nutrition.
  Interventions: Dietary Supplement: enteral nutrition
- parenteral nutrient group (No Intervention)

INTERVENTIONS:
Dietary Supplement: enteral nutrition
  Arms: EN group

SUMMARY:
Different studies suggest that early enteral nutrition (EEN) has benefits in reducing infectious complications, there is no data that addresses whether delayed enteral nutrition (EN) is detrimental and if it may have effects on inflammatory responses and immune function.

ELIGIBILITY:
Inclusion Criteria:

* having a fasting time of more than 14 days
* American Society of Anesthesiologists (ASA) physical status ranging between 1 and 3, and their condition allows enteral nutrition therapy.

Exclusion Criteria:

* chronic renal failure (peritoneal or hemodialysis or creatinine > 2.5 mg/dl)
* history of chronic obstructive pulmonary disease
* hepatic dysfunction or cirrhosis or a bilirubin value > 3 mg/dl
* metabolic diseases,severe anemia
* blood coagulation dysfunction
* pregnancy lactation
* history of psychiatric illness
* patients underwent immunosuppressive therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 28 days

SECONDARY OUTCOMES:
organ failure | 7 days

OTHER OUTCOMES:
inflammatory markers | 7 days
  white blood cell count, C reactive protein(CRP), pro-inflammatory cytokines (TNF-a,IL-1,IL-6), and anti-inflammatory cytokines (IL-4, IL-10)